CLINICAL TRIAL: NCT05122338
Title: Effect of Ultrasound-guided Transversus Abdominis Plane Block With Compound Lidocaine and Esketamine on Postoperative Pain in Patients Undergoing Colorectal Cancer Surgery: a Randomized Double-blind Controlled Trial
Brief Title: Effect of Transversus Abdominis Plane Block With Compound Lidocaine and Esketamine on Pain After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang021
Record Dates: First submitted 2021-11-07; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Pain
Keywords: Compound lidocaine; Ropivacaine; Transversus abdominis plane block; opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution; Sodium Chloride; Ropivacaine; Esketamine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal saline in transversus abdominis plane block (Placebo Comparator): Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side.
  Interventions: Drug: Normal saline
- Ropivacaine in transversus abdominis plane block (Active Comparator): Before the induction of anesthesia, 0.375% ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side.
  Interventions: Drug: Ropivacaine
- Compound lidocaine in transversus abdominis plane block (Active Comparator): Before the induction of anesthesia, 0.4% compound lidocaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side.
  Interventions: Drug: Compound lidocaine
- Compound lidocaine and esketamine in transversus abdominis plane block (Active Comparator): Before the induction of anesthesia, 0.4% compound lidocaine and 0.4mg/kg esketamine are used for bilateral transversus abdominis plane block in a volume of 20 mL of each side.
  Interventions: Drug: Compound lidocaine; Drug: Esketamine

INTERVENTIONS:
Drug: Normal saline — Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: 0. 9% Sodium Chloride Injection
  Arms: Normal saline in transversus abdominis plane block
Drug: Ropivacaine — Before the induction of anesthesia, 0.375% ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Ropivacaine Hydrochloride Injection
  Arms: Ropivacaine in transversus abdominis plane block
Drug: Compound lidocaine — Before the induction of anesthesia, 0.4% compound lidocaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Compound Lidocaine Hydrochloride Injection
  Arms: Compound lidocaine and esketamine in transversus abdominis plane block; Compound lidocaine in transversus abdominis plane block
Drug: Esketamine — Before the induction of anesthesia, 0.4mg/kg esketamine is used for bilateral transversus abdominis plane block
  Other Names: Esketamine injection
  Arms: Compound lidocaine and esketamine in transversus abdominis plane block

SUMMARY:
Purpose:

To explore effects of ultrasound-guided transversus abdominis plane block with compound lidocaine and esketamine on postoperative pain after colorectal cancer surgery.

DETAILED DESCRIPTION:
Poor post-surgical pain control is a leading factor that hinders the physical rehabilitation, and causes acute cognitive impairment and chronic pain syndrome. Recently, the multimodal analgesia strategies to minimise opioid related side effects are highly desirable in open surgical procedures. The transversus abdominis plane block is a novel technique involving injection of local anaesthetic between the internal oblique and the transversus abdominis muscles of the abdominal wall. Although ropivacaine is most commonly used for this technique, the analgesic duration remains not dissatisfied. Compared with ropivacaine, compound lidocaine injection has a better and longer analgesic activity since it contains menthol and ethanol with appropriate concentrations. However, whether compound lidocaine injection is efficiency in the transversus abdominis plane block for abdominal surgery lacks investigations. Herein, we will evaluate the efficacy of ultrasound-guided transversus abdominis plane (USG-TAP) block with compound lidocaine injection and esketamine for postoperative analgesia in patients undergoing colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo colorectal cancer surgery under general anesthesia
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.

Exclusion Criteria:

1. Subject has a diagnosis of bronchial asthma, coronary heart disease, severe hypertension, renal failure or liver failure.
2. Subject has a diagnosis of Insulin dependent diabetes.
3. Subject is allergy and contraindication to local anesthetics or any components of local anesthetics.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre- existing therapy with opioids, intake of any analgesic drug within 48 hours before surgery.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.
7. Subject is obese (body mass index >30kg/m^2).
8. Subject is incapacity to comprehend pain assessment and cognitive assessment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 48 hours after surgery
  Each patient was administered analgesics using a PCA (Patient-controlled analgesia) pump containing opioid in normal saline after leaving PACU (Postanesthesia care unit). Opioid cumulative consumption is recorded for 48 hours postoperatively.

SECONDARY OUTCOMES:
Pain Score (NRS) | 48 hours after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Time of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of opioid.
Total Dose of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of opioid.
The incidence of Side Effects | 48 hours after surgery
  The number of patients with side effects including nausea, vomiting, dizziness, headache, shivering, and pruritus is recorded for 48 hours postoperatively.
Apfel score | The 1 day before the surgery
  The Apfel score was recorded for evaluating risk for developing postoperative nausea and vomiting (PONV).
Mean time until passage of flatus | 96 hours after surgery
  Gastrointestinal motility was evaluated by recording mean time until passage of flatus
Diffusion area of local anesthetics after transversus abdominis plane block | 30 minutes after transversus abdominis plane block
  Diffusion area of local anesthetics after transversus abdominis plane block was calculated under ultrasound assistance.
Normalized Area of Hyperalgesia Around the Incision | 48 hours after surgery
  The skin around the incision is stimulated in steps of 5 mm at intervals of 1 s starting outside of the hyperalgesic area in the direction of the incision. The distance from the incision to the first point where a 'painful', 'sore' or 'sharper'feeling occurred is measured and noted. This measurement is repeated at predefined radial lines around the incision. To eliminate the variable length of incision, this length is subtracted from the longer diameter leaving four radial distances from the end and from the middle of the incision. The normalized area of hyperalgesia is calculated by summing up the areas of the remaining four triangles measured by and Von Frey filament.
The level of cytokines in blood By ELISA kits | 48 hours after surgery
  Blood is collected to measure the level of cytokines (such as IL-18, IL-17, IL-23 ) using ELISA kits.
The level of chemokines in blood By ELISA kits | 48 hours after surgery
  Blood is collected to measure the level of chemokines (such as CXCL1, CCL7, CCL2) using ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, Study Director — Tianjin Medical University General Hospital

IPD SHARING:
Plan to Share IPD: No